CLINICAL TRIAL: NCT01456637
Title: Online Self-Help Intervention for Insomnia: With or Without Feedback
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Utrecht University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPG-20106524
Record Dates: First submitted 2011-10-20; First posted 2011-10-21 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Insomnia
Keywords: Insomnia; Intervention; Self-help; Internet
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT for insomnia with feedback (Experimental): In this arm participants received internet based self-help CBT for insomnia with e-mail feedback form a therapist.
  Interventions: Behavioral: CBT for insomnia
- CBT for insomnia without feedback (Experimental): In this arm participants receive internet based self-help CBT for insomnia without feedback from a therapist.
  Interventions: Behavioral: CBT for insomnia

INTERVENTIONS:
Behavioral: CBT for insomnia — The techniques used throughout the self-help manual are all effective in reducing insomnia: 1) Stimulus control: patients should only go to bed when sleepy, use the bed and bedroom for sleep (and sex) only, maintain a regular rising time, avoid daytime naps and get out of bed and go into another room when unable to fall asleep within 15-20 minutes (return only when sleepy). 2) progressive muscle relaxation. 3) sleep hygiene education (improving health and environmental factors that affect sleep). 3). Sleep restriction, whereby participants will stay only the time in bed that they sleep. 4) cognitive therapy to challenge and dispute incorrect and unhelpful thoughts about sleep (e.g. I must sleep at least 8 hours, otherwise I'll be a wreck tomorrow).

SUMMARY:
The object of this study is to determine whether feedback added to a self-help protocol for insomnia enhances the treatment effect. In this study all participants receive an online self-help cognitive behavioral therapy (CBT) intervention consisting of information (psycho-education) about sleep and cognitive-behavioural exercises. Adult persons with insomnia will be invited via a popular scientific website to fill out online questionnaires. Half of the participants will received by e-mail from a therapist, the other half of the participants will do the intervention without feedback. Participants will be measured 4, 16, and 40 weeks after intervention with the same questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia
* Access to internet
* Dutch citizen

Exclusion Criteria:

* Alcohol or substance abuse
* Being suicidal
* Sleep apnea
* Schizophrenic or having a psychosis disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sleep diary | baseline
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Sleep Quality.
Diary | 4-week follow-up
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Sleep Quality.
Diary | 6 month follow-up
  Daily self-observation used to calculate Total Sleep Time, Wake After Sleep Onset, Sleep Onset Latency, Sleep Efficiency, and Sleep Quality.

SECONDARY OUTCOMES:
Insomnia Severity | baseline
  Insomnia Severity Index
Insomnia severity | 4-week follow-up
  Insomnia Severity Index
Insomnia Severity | 6 month follow-up
  Insomnia Severity Index
Anxiety | baseline
  HADS
Anxiety | 4-week follow-up
  HADS
Anxiety | 6-month follow-up
  HADS
Depression | baseline
  CES-D
Depression | 4-week follow-up
  CES-D
Depression | 6-month follow-up
  CES-D

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Lancee, PhD, Principal Investigator — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Utrecht, Netherlands

REFERENCES:
- See also: Link Text: Popular scientific website about insomnia — http://www.insomnie.nl